CLINICAL TRIAL: NCT06760650
Title: Fluorescein-Induced Acute Kidney Injury in Patients With Diabetes and Chronic Kidney Disease
Brief Title: Fluorescein Angiography in Patients With Diabetes and Chronic Kidney Disease
Acronym: Fluo-AKI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Mabel Aoun, Associate Professor, Saint-Joseph University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CEHDF 2587; Tfem-2025-79 (Other: Faculty of Medicine, Saint Joseph University of Beirut)
Record Dates: First submitted 2024-12-26; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease Stage 4; Chronic Kidney Disease Stage 3B; Chronic Kidney Disease Stage 5; Diabetes Mellitus; Fluorescein Angiography; Acute Kidney Injury
Keywords: Fluorescein Angiography; Acute kidney injury; Chronic kidney disease; Diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Acute Kidney Injury | interventions — Fluorescein Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fluorescein angiography (Experimental): Assessing serum creatinine before and after fluorescein angiography
  Interventions: Diagnostic Test: Fluorescein angiography

INTERVENTIONS:
Diagnostic Test: Fluorescein angiography — Fluorescein angiography
  Other Names: Fluorescein fundus angiography

SUMMARY:
Our study hypothesizes that fluorescein exposure in diabetic patients with advanced chronic kidney disease results in deterioration of kidney function. It will therefore aim to evaluate the incidence of acute kidney injury induced by fluorescein in diabetic patients with CKD. The objective is to determine the incidence, severity and risk factors associated with this deterioration to improve the care of this specific population.

DETAILED DESCRIPTION:
This study will assess the change in serum creatinine in patients with diabetes and advanced chronic kidney disease, after a fluorescein angiography. This is a before and after study that will include 35 patients from the department of ophtalmology over 6 months with a total follow-up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old with type 2 or type 1 diabetes and chronic kidney disease stage 3b to 5 (eGFR<45 mL/min/1.73 m2)

Exclusion Criteria:

* Patients who do not give their consent
* Patients who are allergic to fluorescein
* Patients who are on dialysis
* Patients who had fever, vomiting, diarrhea or any dehydration 48 hours before the intervention
* Patients who had a treatment modification one week before the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-01-07 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Change in serum creatinine | At day 4
  Change in serum creatinine from baseline to day 4

SECONDARY OUTCOMES:
Long-term change in serum creatinine | 3 months
  Change in serum creatinine from baseline to end of the third month

CONTACTS AND LOCATIONS:
Overall Officials: Mabel AOUN, M.D., M.P.H., Principal Investigator — Faculty of Medicine, Saint Joseph University of Beirut
Locations (1):
- Faculty of Medicine, Saint Joseph University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided